CLINICAL TRIAL: NCT04143542
Title: Comparison of Quadratus Lumborum Block 2 and Transversus Abdominis Plan Block for Postoperative Analgesia in Abdominal Surgery
Brief Title: Trunks Body Blocks for Postoperative Analgesia in Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Ceyda Ozhan Caparlar, md, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: QLB 2
Record Dates: First submitted 2019-10-23; First posted 2019-10-29 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Analgesia; Block
Keywords: quadratus lumborum block; transversus abdominis block; postoperative analgesia
MeSH Terms: conditions — Agnosia; Bites and Stings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Groups Q (Experimental): In abdominal surgeries, USG guided Quadratus Lumborum 2 blocks are performed for postoperative analgesia. For this purpose, Quadratus Lumborum Block 2 (QLB 2) are frequently used blocks.
  The aim to this study was to evaluate the postoperative analgesia of preoperative trunk blocks, intraoperative hemodynamic changes with the unblocked control group, Modified Aldrete Recovery Score (MADS) 9 in the recovery unit, Numerical pain scale (NRS) in the service department, It is aimed to examine and compare the time it reaches on the 1st, 2nd and 24th hours after this period. Patient satisfaction is also evaluated in the ward.
  Interventions: Procedure: trunk blocks
- Groups T (Experimental): In abdominal surgeries, USG guided TAP blocks are performed for postoperative analgesia. For this purpose, TAP blocks are frequently used blocks.
  The aim to this study was to evaluate the postoperative analgesia of preoperative trunk blocks, intraoperative hemodynamic changes with the unblocked control group, Modified Aldrete Recovery Score (MADS) 9 in the recovery unit, Numerical pain scale (NRS) in the service department, It is aimed to examine and compare the time it reaches on the 1st, 2nd and 24th hours after this period. Patient satisfaction is also evaluated in the ward.
  Interventions: Procedure: trunk blocks
- Groups C (No Intervention): There was no intervention. All patients will receive pre-oxygenation with O2 100% for 3 min. Anesthesia will be induced by using fentanyl 1μg/kg, propofol 1.5-2 mg/kg, and atracurium 0.5 mg/kg will be used for muscle relaxation. Anesthesia will be maintained by controlled ventilation with oxygen and air (50:50) with the target of EtCO2≈ 35-40 mmHg, isoflurane 1:1.5 minimum alveolar concentration (MAC). Anesthesia will be discontinued and tracheal extubation will be done once the patient fulfills the extubation criteria.Tramadol 100 mg i.v. Before 15 min end of surgery. The patient control analgesia device will administer all patients.

INTERVENTIONS:
Procedure: trunk blocks — Comparison of trunks blocks and control groups for Postoperative Analgesia in Abdominal Surgery
  Arms: Groups Q; Groups T

SUMMARY:
This study aims to the comparison of Quadratus Lumborum Block 2 and Transversus Abdominis Plan Block for Postoperative Analgesia in Abdominal Surgery

DETAILED DESCRIPTION:
This study aims to the comparison of Quadratus Lumborum Block 2 and Transversus Abdominis Plan Block for Postoperative Analgesia in Abdominal Surgery.

In abdominal surgeries, USG guided body blocks are performed for postoperative analgesia. For this purpose, Transversus Abdominis Plan Block (TAPB) and Quadratus Lumborum Block 2 (QLB 2) are frequently used blocks.

The aim of this study was to evaluate for postoperative analgesia of preoperative trunk blocks, intraoperative hemodynamic changes with the unblocked control group, Modified Aldrete Recovery Score (MADS) 9 in the recovery unit, Numerical pain scale (NRS) in the service department, It is aimed to examine and compare the time it reaches on the 1st, 2nd and 24th hours after this period. Patient satisfaction is also evaluated in the ward.

ELIGIBILITY:
Inclusion Criteria:

Abdominal surgery

Exclusion Criteria:

Cardio-respiratory disease Anti-inflammatory treatment Cognitive disorders Written consent form haven't get history of relevant drug allergy infection of the skin at the site of the needle puncture area coagulopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-23 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 1 hours
  The degree of pain will be measured with a numerical rating scale (NRS). All patients' postoperative pain logarithmic rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
Postoperative pain | 2 hours
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
Postoperative pain | 4 hours
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
The degree of postoperative pain | 24 hours
  The degree of pain will be measured with a numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ceyda Ozhan Caparlar, Study Director — Diskapi Yildirim Beyazit Education and Research Hospital